CLINICAL TRIAL: NCT06340139
Title: Additional Effects of Vestibulo-Ocular Reflex Exercises to Improve Balance and Reduce Stimming in Adolescents With Autism Spectrum Disorder.
Brief Title: Vestibulo-Ocular Reflex for Balance and Stimming in Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS-ISB/REC/01742
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (Active Comparator): Conventional treatment group will receive Trampoline jumping, gym ball exercises, sensory diet (joint compressions, deep pressure, head massage) for 4 days a week for 6 weeks
  Interventions: Other: conventional treatment
- Experimental treatment (Experimental): the Vestibulo ocular reflex exercises added with conventional treatment will be given to the second group. Vestibulo-ocular reflex exercises will be performed in phases with phase 1 being a fixation point and phase 2 including head and eye movements. Vestibulo ocular reflex exercises will be started from a 5-minute duration and gradually increased to 60 minutes duration
  Interventions: Other: experimental treatment

INTERVENTIONS:
Other: conventional treatment — conventional treatment with Trampoline jumping, gym ball exercises, sensory diet (joint compressions, deep pressure, head massage
  Arms: Conventional Treatment
Other: experimental treatment — 1 being a fixation point and phase 2 including head and eye movements
  Arms: Experimental treatment

SUMMARY:
Autism spectrum disorder is a neurodevelopmental disorder that encompasses a number of disorders specifically affecting social skills, Communication and present with Rapid repetitive behaviors. Autism spectrum disorder also presents with inability of body to process sensory information which can causes symptoms such as balance deficits, sensitivity to certain sounds or an exaggerated reaction to a normal stimulus. Autism spectrum disorder can affect the quality of life of an individual to a severe extent. This disorder due to sensory processing deficits also shows difficulty in motor planning, coordination and execution of tasks which can make performing activities of daily living highly difficult to perform. It is called a developmental disorder because it affects the growth. Milestones are often delayed in individuals with autism. Due to these deficits individual with autism if not provided with therapies at the right age can stay dependent on caretaker for their whole life. Rapid repetitive behaviors also known as self-stimulatory behaviors are a way to compensate with anxiety, difficulty in processing sensory information and are often used to stimulate themselves to feel calm. Though not a diagnostic symptom autism often still presents with vestibular dysfunction which affects the balance. Several individuals with autism have showed abnormal vestibular ocular reflexes; abnormally long latency of saccades. Rehabilitation protocol of Autism often includes symptomatic treatment and several therapy protocols such as physical therapy, occupational therapy, applied behavior analysis therapy and play therapy.

DETAILED DESCRIPTION:
Stimming behaviors and balance deficits play a huge role in life of an individual with autism. There is indeed a huge gap and lack of literature on how or if exercise protocols from physical therapy can influence balance and reduce stimming behaviors. Although, Previous studies have recommended that Balance and stimming are directly related and that vestibular dysfunction plays a huge role in frequency of stereotyped stimming behaviors. The aim of the study is to investigate the effects of Vestibulo Ocular reflex exercises on balance and frequency of stimming. This study will also influence how a physical therapist can improve quality of life of an individual with autism by reducing their stimming behavior. Earlier studies also mentioned that Vestibular ocular reflex is affected in kids with autism. Hence this study can play an important role in determining the direct connection between these behaviors, Vestibular ocular reflex and balance.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-18 years
* Both male and female
* Diagnosed Autism Spectrum disorder.
* Visual and/or Vestibular stimming diagnosed by physician.

Exclusion Criteria:

* Patients diagnosed with other neurological diseases
* Tumors or neoplasms
* Visual and auditory impairments
* Inability to respond to verbal command through verbal or non-verbal communication cues.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Aberrant behavior checklist | week 6
  Widely used to assess treatment effects in individuals with developmental disabilities. - Assess emotional and behavioral problems. -
  Consists of 58 items categorized into 5 subscales:
  social withdrawal, irritability, stereotypic behavior,
Berg Balance Scale (BBS) | week 6
  It is often used to assess balance and mobility as well as identify people who are at risk of falling. 14 different balance-related tasks, including sitting, standing, and transferring, are included in the tool. Each factor is scored from 0 to 4, with 0 suggesting significant impairment and 4 denoting the patient's balance system operating normally
Repetitive Behavior Scale - Revised | week 6
  Structured and standardized tool for assessing and characterizing repetitive behaviors in individuals with ASD. - Consists of six subscales: Stereotyped Behavior, Self- Injurious Behavior, Compulsive Behavior, Routine Behavior, Sameness Behavior, and Restricted nterests. - Uses a Likert scale for rating frequency and intensity (0 to 3).
Functional Reach Test | week 6
  A static balance test called the functional reach test is frequently used to evaluate a subject's level of balance when they are standing.The reach distance during this has been used as a measurement for determining fall risk

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afridi, PhD*, Principal Investigator — Riphah International University
Locations (1):
- zamam autism Centre, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No